CLINICAL TRIAL: NCT03001310
Title: An Open Label, Multi-centre, Phase I/II Dose Escalation Trial of a Recombinant Adeno-associated Virus Vector (AAV2/8-hCARp.hCNGB3) for Gene Therapy of Adults and Children With Achromatopsia Owing to Defects in CNGB3
Brief Title: Gene Therapy for Achromatopsia (CNGB3)
Acronym: CNGB3
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MeiraGTx UK II Ltd (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MGT006; 2016-002290-35 (EudraCT Number)
Record Dates: First submitted 2016-11-22; First posted 2016-12-23 (Estimated); Results first posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Achromatopsia
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Biological-Low dose AAV - CNGB3 (Experimental): Subretinal administration of a single low dose of AAV - CNGB3
  Interventions: Biological: AAV - CNGB3
- Biological-Medium dose AAV - CNGB3 (Experimental): Subretinal administration of a single intermediate dose of AAV - CNGB3
  Interventions: Biological: AAV - CNGB3
- Biological-High dose AAV - CNGB3 (Experimental): Subretinal administration of a single high dose of AAV - CNGB3
  Interventions: Biological: AAV - CNGB3

INTERVENTIONS:
Biological: AAV - CNGB3 — Comparison of different dosages of AAV-CNGB3

SUMMARY:
A clinical trial of AAV - CNGB3 retinal gene therapy for patients with achromatopsia

DETAILED DESCRIPTION:
CNGB3 retinal gene therapy for patients with achromatopsia

ELIGIBILITY:
Inclusion Criteria:

* Are aged 3 years or older
* Have achromatopsia confirmed by a retinal specialist (CI or PI)

Exclusion Criteria:

* Are females who are pregnant or breastfeeding
* Have participated in another research study involving an investigational medicinal therapy for ocular disease within the last 6 months
* Have any other condition that the CI/PI considers makes them inappropriate for entry into the trial

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Bainbridge, Prof, Principal Investigator — Chief Investigator
Locations (2):
- University of Michigan Kellog Eye Centre, Ann Arbor, Michigan, United States
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michaelides M, Hirji N, Wong SC, Besirli CG, Zaman S, Kumaran N, Georgiadis A, Smith AJ, Ripamonti C, Gottlob I, Robson AG, Thiadens A, Henderson RH, Fleck P, Anglade E, Dong X, Capuano G, Lu W, Berry P, Kane T, Naylor S, Georgiou M, Kalitzeos A, Ali RR, Forbes A, Bainbridge J. First-in-Human Gene Therapy Trial of AAV8-hCARp.hCNGB3 in Adults and Children With CNGB3-associated Achromatopsia. Am J Ophthalmol. 2023 Sep;253:243-251. doi: 10.1016/j.ajo.2023.05.009. Epub 2023 May 11. PMID 37172884

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from medical centers in the United Kingdom (UK) and the United States (US). A total of 23 participants were enrolled in the study.
Groups:
- Low Dose AAV - CNGB3: Subretinal administration of a single low dose of adeno-associated virus AAV-CNGB3; AAV-CNGB3: AAV gene therapy for defects in CNGB3 gene
- Intermediate Dose AAV-CNGB3: Subretinal administration of a single intermediate dose of adeno-associated virus AAV-CNGB3; AAV-CNGB3: AAV gene therapy for defects in CNGB3 gene
- Other Dose - AAV - CNGB3: Subretinal administration of a single other dose (between intermediate and high dose levels) of adeno-associated virus AAV-CNGB3; AAV-CNGB3: AAV gene therapy for defects in CNGB3 gene
- High Dose AAV - CNGB3: Subretinal administration of a single high dose of adeno-associated virus AAV-CNGB3; AAV-CNGB3: AAV gene therapy for defects in CNGB3 gene
Period: Overall Study
Arm/Group | Low Dose AAV - CNGB3 | Intermediate Dose AAV-CNGB3 | Other Dose - AAV - CNGB3 | High Dose AAV - CNGB3
Started | 3 | 12 | 3 | 5
Completed | 3 | 12 | 3 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose AAV - CNGB3 | Intermediate Dose AAV-CNGB3 | Other Dose - AAV - CNGB3 | High Dose AAV - CNGB3 | Total
Number analyzed (Participants) | 3 | 12 | 3 | 5 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 8 | 3 | 2 | 13
  Between 18 and 65 years | 3 | 4 | 0 | 3 | 10
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 3 | 3 | 18
  Male | 1 | 2 | 0 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 12 | 3 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 12 | 3 | 5 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 0 | 1 | 2 | 0 | 3
  United Kingdom | 3 | 11 | 1 | 5 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting the Primary Outcome Defined as Any of the Below Events Occurring During the 6 Weeks Following Administration, at Least Possibly Related to the Advanced Therapy Investigational Medicinal Products (ATIMP), Not Surgery Alone.
Description: The primary outcome is defined as any of the below occurring during the 6 weeks following administration, at least possibly related to the Advanced Therapy Investigational Medicinal Products (ATIMP), not surgery alone:
  * Reduction in visual acuity by 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters or more that fails to resolve to within 15 letters of baseline in a 4-week period once prophylactic treatment commences
  * Severe unresponsive inflammation
  * Infective endophthalmitis
  * Ocular malignancy
  * Grade III or above non-ocular Suspected Unexpected Serious Adverse Reaction (SUSAR)
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose AAV - CNGB3 | Intermediate Dose AAV-CNGB3 | Other Dose - AAV - CNGB3 | High Dose AAV - CNGB3
Number analyzed (Participants) | 3 | 12 | 3 | 5
Participants | 0 | 1 | 0 | 2

2. Secondary Outcome: Improvements in Visual Function as Assessed by Visual Acuity
Description: Change from baseline to Week 24 in best corrected visual acuity (BCVA) using Early Treatment Diabetic Retinopathy Study (ETDRS) chart letter score in the treated eye. The direction of improvement from baseline is an increase in the number of ETDRS letters read over time.
Time Frame: 6 months
Population: 22 of the 23 participants performed the visual acuity assessment at baseline and Week 24.
Measure: Mean (Full Range); unit: number of ETDRS letters
Arm/Group | Low Dose AAV - CNGB3 | Intermediate Dose AAV-CNGB3 | Other Dose - AAV - CNGB3 | High Dose AAV - CNGB3
Number analyzed (Participants) | 3 | 11 | 3 | 5
number of ETDRS letters | -0.44 [-2.0 to 1.3] | -0.58 [-4.3 to 3.3] | 1.78 [0.3 to 4.7] | 1.45 [-4.0 to 5.3]

3. Secondary Outcome: Improvements in Retinal Function as Assessed by Static Perimetry
Description: Change from baseline to Week 24 in mean retinal sensitivity in the treated eye. The direction of improvement is an increase in sensitivity.
Time Frame: 6 months
Population: 20 of the 23 participants had mean retinal sensitivity data available at both baseline and Week 24 in the treated eye.
Measure: Mean (Full Range); unit: decibel
Arm/Group | Low Dose AAV - CNGB3 | Intermediate Dose AAV-CNGB3 | Other Dose - AAV - CNGB3 | High Dose AAV - CNGB3
Number analyzed (Participants) | 3 | 9 | 3 | 5
decibel | -1.58 [-3.1 to 0.0] | -0.39 [-2.4 to 1.8] | 8.13 [1.7 to 11.4] | -0.77 [-7.1 to 3.3]

4. Secondary Outcome: Quality of Life Measured by QoL Questionnaires in Children and Adolescents
Description: Change from baseline to Week 24 in EuroQol-5D-Y Visual Analogue Scale (EQ-VAS) in children and adolescents. EQ-VAS uses a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. A positive change from baseline reflects improvement and a negative change from baseline reflects worsening.
Time Frame: 6 months
Population: EQ-VAS data were available for 11 children/adolescents enrolled in the study.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Low Dose AAV - CNGB3 | Intermediate Dose AAV-CNGB3 | Other Dose - AAV - CNGB3 | High Dose AAV - CNGB3
Number analyzed (Participants) | 0 | 7 | 3 | 1
units on a scale |  | 6.9 [-2 to 20] | 2.3 [-3 to 10] | -9.0

5. Secondary Outcome: Quality of Life Measured by QoL Questionnaires in Adults
Description: Change from baseline to Week 24 in EuroQol-5D-5L Visual Analogue Scale (EQ-VAS) in adults. EQ-VAS uses a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state. A positive change from baseline reflects improvement and a negative change from baseline reflects worsening.
Time Frame: 6 Months
Population: EQ-VAS data were available for 11 adults enrolled in the study.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Low Dose AAV - CNGB3 | Intermediate Dose AAV-CNGB3 | Other Dose - AAV - CNGB3 | High Dose AAV - CNGB3
Number analyzed (Participants) | 3 | 4 | 0 | 4
units on a scale | 0.0 [-10 to 10] | -3.8 [-10 to 5] |  | 4.3 [-5 to 20]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Total: Safety Analysis Set
Arm/Group | Low Dose AAV - CNGB3 | Intermediate Dose AAV-CNGB3 | Other Dose - AAV - CNGB3 | High Dose AAV - CNGB3 | Total
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/12 | 0/3 | 0/5 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/12 | 0/3 | 1/5 | 2/23
Other Adverse Events (participants affected / at risk) | 3/3 | 12/12 | 3/3 | 5/5 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose AAV - CNGB3 (N=3) | Intermediate Dose AAV-CNGB3 (N=12) | Other Dose - AAV - CNGB3 (N=3) | High Dose AAV - CNGB3 (N=5) | Total (N=23)
Uveitis (Eye disorders) | 0 | 1 | 0 | 1 | 2
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose AAV - CNGB3 (N=3) | Intermediate Dose AAV-CNGB3 (N=12) | Other Dose - AAV - CNGB3 (N=3) | High Dose AAV - CNGB3 (N=5) | Total (N=23)
Conjunctival haemorrhage (Eye disorders) | 3 | 10 | 2 | 5 | 20
Lenticular opacities (Eye disorders) | 2 | 7 | 3 | 3 | 15
Visual acuity reduced (Eye disorders) | 2 | 7 | 1 | 5 | 15
Subretinal fluid (Eye disorders) | 2 | 4 | 0 | 3 | 9
Foreign body sensation in eyes (Eye disorders) | 0 | 7 | 0 | 1 | 8
Ocular discomfort (Eye disorders) | 0 | 5 | 0 | 3 | 8
Chorioretinal folds (Eye disorders) | 0 | 4 | 0 | 2 | 6
Retinal haemorrhage (Eye disorders) | 2 | 2 | 0 | 2 | 6
Conjunctival hyperaemia (Eye disorders) | 0 | 3 | 1 | 0 | 4
Eye inflammation (Eye disorders) | 1 | 1 | 2 | 0 | 4
Maculopathy (Eye disorders) | 0 | 1 | 0 | 3 | 4
Retinal depigmentation (Eye disorders) | 0 | 2 | 2 | 0 | 4
Retinal oedema (Eye disorders) | 0 | 2 | 0 | 2 | 4
Retinal tear (Eye disorders) | 0 | 3 | 0 | 1 | 4
Eye pain (Eye disorders) | 0 | 2 | 1 | 0 | 3
Photophobia (Eye disorders) | 0 | 2 | 0 | 1 | 3
Vitreous floaters (Eye disorders) | 1 | 2 | 0 | 0 | 3
Conjunctival oedema (Eye disorders) | 0 | 2 | 0 | 0 | 2
Corneal disorder (Eye disorders) | 0 | 1 | 0 | 1 | 2
Macular fibrosis (Eye disorders) | 0 | 1 | 0 | 1 | 2
Retinal disorder (Eye disorders) | 0 | 1 | 1 | 0 | 2
Retinal pigment epitheliopathy (Eye disorders) | 0 | 2 | 0 | 0 | 2
Uveitis (Eye disorders) | 0 | 0 | 0 | 2 | 2
Headache (Nervous system disorders) | 1 | 3 | 1 | 1 | 6
Visual field defect (Nervous system disorders) | 0 | 4 | 0 | 1 | 5
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 1 | 4
Rhinitis (Infections and infestations) | 0 | 4 | 0 | 1 | 5
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2
Intraocular pressure increased (Investigations) | 2 | 1 | 1 | 2 | 6
Fatigue (General disorders) | 0 | 2 | 0 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT03001310/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT03001310/SAP_001.pdf